CLINICAL TRIAL: NCT06607731
Title: Percutaneous Gelled Alcohol Sclerotherapy for Aggressive Angiomas: Evaluation of Feasibility, Safety, and Efficacy
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN312024/CHUSTE
Record Dates: First submitted 2024-07-26; First posted 2024-09-23 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Bone Angioma
Keywords: percutaneous sclerosis; ethanol gel; aggressive bone angioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Patients who have undergone percutaneous gel ethanol sclerosis for aggressive bone angioma at Saint-Etienne University Hospital.
  Interventions: Other: Collecting data from medical records

INTERVENTIONS:
Other: Collecting data from medical records — Data collected: clinical data (particularly pain), biological data, imaging.

SUMMARY:
The investigators aimed to evaluate efficacy and safety of a non-surgical protocol treatment combining transarterial embolization and percutaneous radiopaque gelled ethanol (RGE) sclerotherapy in a first procedure, then followed by vertebroplasty in a second procedure, to treat aggressive vertebral hemangioma patients in tertiary hospital. Exclusion criteria were age <18-years old and any association with neurological deficit.

ELIGIBILITY:
Inclusion Criteria:

* Every patients treated by gelled alcohol sclerotherapy for aggressive angiomas, in the University Hospital of Saint-Etienne.

Exclusion Criteria:

* Patients no treated by gelled alcohol sclerotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent percutaneous gel ethanol sclerosis for aggressive bone angioma at Saint-Étienne University Hospital will be included.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of complications identified in data collection | Day 1
  Number of complications identified in data collection

SECONDARY OUTCOMES:
Number of lesion identified in data collection | Day 1
  Number of lesion identified in data collection

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain GRANGE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Priest-en-Jarez, France

IPD SHARING:
Plan to Share IPD: No